CLINICAL TRIAL: NCT02185885
Title: The Importance of Mean Arterial Pressure During Cardiopulmonary Bypass to Prevent Cerebral Complications After Cardiac Surgery - a Randomised Clinical Trial.
Brief Title: Perfusion Pressure Cerebral Infarction Trial (PPCI)
Acronym: PPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Jens C. Nilsson, Consultant, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-3-2013-110; E-22329-01 (Other: Rigshospitalet, project.no.); 4142, PPCI (Other: Dep. of Cardiothoracic Anesthesiology)
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Embolic Stroke; Postoperative Cognitive Dysfunction
Keywords: Ischemic stroke; Embolic stroke; Postoperative Cognitive Dysfunction; Cardiac Bypass Surgery; Cardiac Anaesthesia
MeSH Terms: conditions — Embolic Stroke; Postoperative Cognitive Complications; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased bloodpressure during CPB (Experimental): The cardiopulmonary bypass (CPB) procedure is conducted according to department guidelines with the modification that MAP is kept between 70 and 80 mm Hg. This is achieved by refract intravenous doses of phenylephrine to a total maximum of 2.0 mg, and after that continuous intravenous infusion of norepinephrine up to 0.4 μg/kg/min if necessary.
  Interventions: Procedure: Increased bloodpressure during CPB.
- Regular bloodpressure during CPB (No Intervention): The cardiopulmonary bypass (CPB) procedure is conducted in accordance with departmental guidelines, where MAP is sought to be ≥ 45 mm Hg. This is achieved by refract intravenous doses of phenylephrine to a total maximum of 2.0 mg, and after that continuous intravenous infusion of norepinephrine up to 0.4 μg/kg/min if necessary.

INTERVENTIONS:
Procedure: Increased bloodpressure during CPB.
  Arms: Increased bloodpressure during CPB

SUMMARY:
STUDY HYPOTHESIS

In cardiac surgery the volume of perioperative cerebral infarctions can be reduced by increasing mean arterial pressure (MAP) during the cardiopulmonary bypass procedure.

BRIEF STUDY SUMMARY

Heart surgery using cardiopulmonary bypass (CPB) can be complicated by injury to the brain. Previous studies using brain scans have reported small stroke-like lesions in up to 51% of patients after cardiac surgery. However, only 1-6 % of patients have permanent symptoms of severe brain damage.

The majority of brain lesions seem to be caused by particulate matter (emboli) that wedge in blood vessels of the brain thereby compromising flow. In addition, insufficient blood flow to areas of the brain supplied by narrowed, calcified vessels may contribute. MAP during CPB usually stabilizes below the lower limit of cerebral autoregulation, which is accepted since sufficient total blood flow is guaranteed during CPB.

The aim of the PPCI trial is to investigate if increased MAP during CPB can prevent or reduce the extent of brain injury after cardiac surgery. A beneficial effect could result from reduced embolic injury through increased blood flow in collateral vessels and/or by increased blood flow in calcified arteries.

180 patients scheduled for cardiac surgery will be randomly allocated to increased MAP (70-80 mm Hg) or 'usual practice' (typically 45-50 mm Hg) during CPB, whereas CPB blood flow is intended equal and fixed in the two groups. Patients are examined before and 3-6 days after surgery with magnetic resonance imaging (MRI) brain scans, mental tests and by blood borne markers of brain injury.

If higher MAP during CPB is beneficial, a change of practice can easily be implemented in the clinical routine.

DETAILED DESCRIPTION:
TRIAL DESIGN

The PPCI trial is a randomized, controlled, outcomes assessor and patient blinded, single-center superiority trial with two parallel groups in a 1:1 allocation ratio. The randomization will be stratified according to age (stratum 1 < 70 years; stratum 2 ≥ 70 years) and type of surgery (stratum 1 - surgery involving the aortic and/or mitral valve; stratum 2 - surgery not involving these valves).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* scheduled elective or subacute cardiac surgery with the use of CPB.
* type of surgery either coronary artery bypass grafting (CABG) and/or heart valve surgery (provided that the valve prosthesis used is MRI compatible).

Exclusion Criteria:

* a history of stroke.
* a history of reversible ischemic deficits (duration of symptoms 24-72 hours)
* a history of transitory ischemic attacks (duration of symptoms < 24 hours)
* diagnosis of neurodegenerative disorders such as Alzheimers, Multiple Sclerosis etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Total volume of new ischemic cerebral lesions | 6 days
  The total volume of new ischemic cerebral lesions (sum in mL) assessed by diffusion-weighed-magnetic resonance imaging conducted preoperatively and again once postoperatively on day 3 to 6.
  The analysis will be adjusted for the randomization stratification variables age and type of surgery.

SECONDARY OUTCOMES:
Total number of new ischemic cerebral lesions | 6 days
  The total number of new ischemic cerebral lesions (sum in mL) assessed by diffusion-weighed-magnetic resonance imaging conducted preoperatively and again once postoperatively on day 3 to 6.
Magnetic resonance spectroscopy - change from baseline N-acetylaspartate-creatine (NAA/Cr) ratio at day 6 | 6 days
  Diffuse cerebral injury is investigated using Single-Voxel Magnetic Resonance Spectroscopy (MRS) in grey and white cerebral matter and expressed as the difference in N-acetylaspartate-creatine (NAA/Cr) ratio between a scan conducted preoperatively and one conducted postoperatively on day 3 to 6.
Magnetic resonance spectroscopy - change from baseline MRS Choline-creatine (Cho/Cr ratio) at day 6 | 6 days
  Diffuse cerebral injury is investigated using Single-Voxel Magnetic Resonance Spectroscopy (MRS) in grey and white cerebral matter and expressed as the difference in Choline-creatine (Cho/Cr ratio) between a scan conducted preoperatively and one conducted postoperatively on day 3 to 6.
Postoperative cognitive dysfunction (POCD) - change from baseline neuropsychological test performance at day 5-8 | 5-8 days
  The presence of cognitive dysfunction is evaluated preoperatively and on day 5-8 using the following collection of specific tests each time: "Visual Verbal Learning test", "Concept Shifting test", "Stroop Colour Word Interference test" and "Letter Digit Coding test".
  Cognitive dysfunction is defined as a deterioration corresponding to a Z-score > 2 (as defined by the ISPOCD group).
Postoperative cognitive dysfunction (POCD) - change from baseline neuropsychological test performance at 3 months | 3 months
  The presence of cognitive dysfunction is evaluated preoperatively and 3 months postoperatively using the following collection of specific tests each time: "Visual Verbal Learning test", "Concept Shifting test", "Stroop Colour Word Interference test" and "Letter Digit Coding test".
  Cognitive dysfunction is defined as a deterioration corresponding to a Z-score > 2 (as defined by the ISPOCD group).
Peak value of biochemical markers of brain injury | Prior to surgery on day 1 and 24 hours, 48 hours and 6 days after surgery
  Blood samples will be drawn at 4 different time points during the admission. Serum concentration and time course of the following markers of brain injury will be assessed: Phosphorylated Neurofilament Heavy Protein (pNfH), Glial Fibrillary Acidic Protein (GFAP), Matrix Metallopeptidase 9 (MMP-9) and Ubiquitin C-terminal Hydrolase 1 (UCH-L1).
Near Infrared Spectroscopy (NIRS) - lowest value | End of surgery
  Near Infrared Spectroscopy (NIRS) NIRS values from the right and left frontal lobes of the brain will be continuously monitored during the intraoperative period and saved for later analysis. The NIRS monitor will be hidden and muted during the procedure.
Near Infrared Spectroscopy (NIRS) - total time below 25% of the baseline value on right and left side | End of surgery
  Near Infrared Spectroscopy (NIRS) NIRS values from the right and left frontal lobes of the brain will be continuously monitored during the intraoperative period and saved for later analysis. The NIRS monitor will be hidden and muted during the procedure.
Change from baseline performance at neurological examination day 6 | 6 days
  New neurological deficits are assessed by performing an objective, clinical neurological examination.

OTHER OUTCOMES:
GAMPT BCC200 count | End of cardiopulmonary bypass procedure
  The GAMPT BCC200 is integrated into the heart-lung-machine (HLM), and through the use of ultrasound Doppler techniques, detection of gaseous micro-emboli (GME, volume between 5-500 µl) is enabled. The system can be used to quantify the GME that pass from the HLM into the bloodstream of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jens C. Nilsson, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Hanne B. Ravn, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiothoracic Surgery 2152 and Department of Cardiothoracic Anesthesiology 4142, Rigshospitalet / Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Derived] Vedel AG, Holmgaard F, Danielsen ER, Langkilde A, Paulson OB, Ravn HB, Rasmussen LS, Nilsson JC. Blood pressure and brain injury in cardiac surgery: a secondary analysis of a randomized trial. Eur J Cardiothorac Surg. 2020 Nov 1;58(5):1035-1044. doi: 10.1093/ejcts/ezaa216. PMID 32840297
- [Derived] Holmgaard F, Vedel AG, Rasmussen LS, Paulson OB, Nilsson JC, Ravn HB. The association between postoperative cognitive dysfunction and cerebral oximetry during cardiac surgery: a secondary analysis of a randomised trial. Br J Anaesth. 2019 Aug;123(2):196-205. doi: 10.1016/j.bja.2019.03.045. Epub 2019 May 17. PMID 31104758
- [Derived] Holmgaard F, Vedel AG, Lange T, Nilsson JC, Ravn HB. Impact of 2 Distinct Levels of Mean Arterial Pressure on Near-Infrared Spectroscopy During Cardiac Surgery: Secondary Outcome From a Randomized Clinical Trial. Anesth Analg. 2019 Jun;128(6):1081-1088. doi: 10.1213/ANE.0000000000003418. PMID 31094772
- [Derived] Holmgaard F, Vedel AG, Langkilde A, Lange T, Nilsson JC, Ravn HB. Differences in regional cerebral oximetry during cardiac surgery for patients with or without postoperative cerebral ischaemic lesions evaluated by magnetic resonance imaging. Br J Anaesth. 2018 Dec;121(6):1203-1211. doi: 10.1016/j.bja.2018.05.074. Epub 2018 Jul 26. PMID 30442245
- [Derived] Vedel AG, Holmgaard F, Rasmussen LS, Langkilde A, Paulson OB, Lange T, Thomsen C, Olsen PS, Ravn HB, Nilsson JC. High-Target Versus Low-Target Blood Pressure Management During Cardiopulmonary Bypass to Prevent Cerebral Injury in Cardiac Surgery Patients: A Randomized Controlled Trial. Circulation. 2018 Apr 24;137(17):1770-1780. doi: 10.1161/CIRCULATIONAHA.117.030308. Epub 2018 Jan 16. PMID 29339351
- [Derived] Vedel AG, Holmgaard F, Rasmussen LS, Paulson OB, Thomsen C, Danielsen ER, Langkilde A, Goetze JP, Lange T, Ravn HB, Nilsson JC. Perfusion Pressure Cerebral Infarct (PPCI) trial - the importance of mean arterial pressure during cardiopulmonary bypass to prevent cerebral complications after cardiac surgery: study protocol for a randomised controlled trial. Trials. 2016 May 17;17(1):247. doi: 10.1186/s13063-016-1373-6. PMID 27189028